CLINICAL TRIAL: NCT03486665
Title: Characterization and Quantitative Analysis of White Blood Cells in the Blood and Cerebrospinal Fluid of MS Patients
Brief Title: Characterization of White Blood Cells Sub-populations From Multiple Sclerosis Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bioimmunate (Industry)
Responsible Party: Sponsor
Other Study IDs: BIT-001
Record Dates: First submitted 2018-03-21; First posted 2018-04-03 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diagnosed with Multiple Sclerosis: Patients previously diagnosed with Multiple Sclerosis
  Interventions: Other: Blood Sampling
- Newly Diagnosed with Multiple Sclerosis: Patients diagnosed for the first time with Multiple Sclerosis and hospitalized
  Interventions: Other: Blood Sampling; Other: CSF Sampling
- Healthy Volunteers: Health volunteers who do not have an autoimmune diseases, including Multiple Sclerosis
  Interventions: Other: Blood Sampling

INTERVENTIONS:
Other: Blood Sampling — Blood samples will be taken from all patients and healthy volunteers.
Other: CSF Sampling — CSF sample will be taken from hospitalized newly diagnosed patients only.
  Groups: Newly Diagnosed with Multiple Sclerosis

SUMMARY:
Multiple sclerosis (MS) is a chronic progressive neurological autoimmune disease, that gradually affects patient's quality of life. There are about 2.5 millions patients world wide, with an increasing cost Burdon. Up to date, it remains unclear who are the exact cells to initiate the disease. During the disease, the repertoire of cells expands and undergoes changes. The purpose of this study is to characterize those changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of MS according to the revised criteria of McDonald or healthy volunteers
* Ability to provide written informed consent.

Exclusion Criteria:

- Active malignant disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 to 70 years old patients with MS defined according to the revised diagnostic criteria of MacDonald and are followed by the neurology or physical medicine and rehabilitation center or healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Quantification of disease related white blood cells from blood and/ or CSF | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel